CLINICAL TRIAL: NCT03655405
Title: Opportunities and Limits to Deprescribing in Nursing Homes: Randomised, Controlled Trial of an Individual Deprescribing Intervention for Nursing Homes Residents.
Brief Title: Randomised, Controlled Trial of an Individual Deprescribing Intervention for Nursing Homes Residents
Acronym: OLD-NH-IDeI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Niquille (Other)
Responsible Party: Sponsor-Investigator, Anne Niquille, Doctor, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OLD-NH-IDeI-2018
Record Dates: First submitted 2018-08-30; First posted 2018-08-31 (Actual); Results first posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Polypharmacy; Inappropriate Prescribing
Keywords: Deprescribing; Nursing Home; Potentially Inappropriate Medication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Deprescribing Intervention (Experimental): Participants allocated to the intervention arm will receive the Individual Deprescribing Intervention (pharmacist-led medication review, followed by the creation of a deprescribing plan by the pharmacist, physician and responsible nurse).
  Interventions: Other: Individual Deprescribing Intervention
- Control (No Intervention): Participants allocated to the control group will receive usual care.

INTERVENTIONS:
Other: Individual Deprescribing Intervention — The pharmacist responsible for the nursing home will perform a medication review (type 3). The results of this review will be discussed with the physician and nurse responsible for this participant, with the goal of creating a personalised deprescribing plan. Once validated by the physician, this plan will be submitted to the participant for approval.
  Arms: Individual Deprescribing Intervention

SUMMARY:
This study will evaluate the effects of a pharmacist-led, deprescribing-focused medication review on the use of inappropriate medications by nursing home residents

DETAILED DESCRIPTION:
Nursing home residents are often prescribed inappropriate medication, drugs whose negative effects outweigh potential benefits or which are not useful anymore. Inappropriate medication have been linked with worse health outcomes, hospitalisations and death. Deprescribing, the structured process of withdrawing or tapering inappropriate medications, has been studied as a potential solution to this problem.

In this study, nursing home residents living in institution which are already engaged in a deprescribing process will be randomly allocated to receive a medication review or usual care. The medication review will be performed by the nursing home pharmacist an its results will be discussed with the responsible physicians and nurses to create a deprescribing plan specifically tailored to the needs of the resident.

ELIGIBILITY:
Inclusion Criteria:

* Take 5 or more prescribed drugs daily;
* Reside in the Nursing Home since at least 4 months.

Exclusion Criteria:

* Physician judges that discussing deprescribing with them risks destabilising them.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bugnon, Prof, Study Director — ISPSO, Universties of Geneva and Lausanne, Switzerland
Locations (1):
- Centre de Pharmacie Communautaire, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Data are available from the investigators upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: 10-year availability
Access Criteria: Data are available from the investigators upon reasonable request.

REFERENCES:
- [Derived] Cateau D, Ballabeni P, Mena S, Bugnon O, Niquille A. Deprescribing in nursing homes: Protocol for nested, randomised controlled hybrid trials of deprescribing interventions. Res Social Adm Pharm. 2021 Apr;17(4):786-794. doi: 10.1016/j.sapharm.2020.05.026. Epub 2020 May 27. PMID 32622774
- See also: Project description on the funding body website — http://www.nfp74.ch/fr/projets/soins-stationnaires/projet-bugnon

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individual Deprescribing Intervention | Control
Started | 32 | 30
Completed | 27 | 25
Not Completed | 5 | 5
Not completed — Death after initial data collection | 4 | 2
Not completed — Died before initial data collection | 1 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intervention: 1 participant excluded, died before initial data collection; Control: 3 participants excluded: 2 died before initial data collection, no data was collected on one.
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Deprescribing Intervention | Control | Total
Number analyzed (Participants) | 31 | 27 | 58
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 87 [80 to 91] | 84 [78 to 88] | 87 [80 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 15 | 7 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 31 | 27 | 58
Duration of stay in years [Mean (Standard Deviation); unit: years] | 3.1 (2.3) | 3.6 (3.6) | 3.4 (2.9)
Number of drugs prescribed [Median (Inter-Quartile Range); unit: drugs] | 15 [12 to 19] | 15 [13 to 18] | 15 [12 to 19]
Number of chronic drugs [Median (Inter-Quartile Range); unit: drugs] | 12 [10 to 14] | 11 [8 to 12] | 11 [9 to 13]
Number of PIMs [Median (Inter-Quartile Range); unit: potentially inappropriate medications] — Number of Potentially Inappropriate Medications (PIMs); appropriateness is assessed using the French translation of the Screening Tool of Older People's Prescription (STOPP) v2.
  potentially inappropriate medications | 5 [4 to 7] | 6 [3 to 7] | 5 [3 to 7]
Number of chronic DDDs [Mean (Standard Deviation); unit: chronic DDD] — Number of chronic Defined Daily Dose (DDD); chronicity is defined as the absence of a planned cessation date in the participant's record. DDDs are assigned according the the World Health Organization's (WHO) DDD set.
  chronic DDD | 9.6 (3.5) | 9.3 (3.6) | 9.5 (4.1)
Number of PIM DDDs [Mean (Standard Deviation); unit: PIM DDD] — Sum of potentially inappropriate DDDs; appropriateness is assessed using the French translation of STOPP v2; DDDs are assigned according to the WHO's DDD set.
  PIM DDD | 3.6 (2.8) | 3.4 (2.1) | 3.5 (2.5)
Quality of life: EQ-5D-5L analog scale [Mean (Standard Deviation); unit: analog scale units] — The EuroQol 5-Dimensions 5-Levels (EQ-5D-5L) tool was used to assess quality of life; this tool includes a visual analog scale, ranging from 0 to 100, 100 indicating "the best health you can imagine" and 0 "the worst health you can imagine". Higher results indicate an higher quality of life.
  analog scale units | 56.5 (24.8) | 61.4 (20.5) | 58.9 (22.8)
Quality of life: EQ-5D-5L index [Mean (Standard Deviation); unit: index] — The quality of life was assessed using EQ-5D-5L; this tool includes 5 questions, each with 5 possible answers. Using a valuation set, the answers to individual questions were transformed in a numeric index value for each participants, with a maximum of 1 and an infinitely low minimum. Higher values indicates higher perceived health-related quality of life.
  index | 0.46 (0.34) | 0.50 (0.33) | 0.48 (0.34)

OUTCOME MEASURES:

1. Primary Outcome: Number of Inappropriate Medication at Follow-up
Description: Number of inappropriate medications prescribed at follow-up, assessed using the French translation of STOPP v2.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: drugs
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
drugs | 4.35 (2.72) | 4.85 (2.58)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.723, Regression, Poisson; Number of PIMs at follow-up, adjusted for baseline value; Incidence Rate Ratio = 0.972, 95% CI 2-sided [0.830 to 1.138]

2. Secondary Outcome: Number of Potentially Inappropriate DDDs Prescribed to Participants at Follow-up
Description: Appropriateness assessed using the French translation of STOPP v2; DDD defined by WHO.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: DDD
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
DDD | 2.73 (2.97) | 3.10 (1.99)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.033, Regression, Poisson; Number of potentially inappropriate DDD at follow-up, adjusted for baseline value; Incidence Rate Ratio = 0.763, 95% CI 2-sided [0.594 to 0.979]

3. Secondary Outcome: Number of Chronic Drugs Prescribed to Participants
Description: Number of Chronic Drugs Prescribed to Participants
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: drugs
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
drugs | 9.68 (3.59) | 9.67 (3.10)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.064, Regression, Poisson; Number of chronic drugs at follow-up, adjusted for baseline value; Incidence Rate Ratio = 0.915, 95% CI 2-sided [0.834 to 1.005]

4. Secondary Outcome: Number of Chronic DDDs Prescribed to Participants
Description: Number of chronic DDDs prescribed to participants
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: DDD
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
DDD | 7.82 (3.85) | 7.65 (2.74)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.857, Regression, Poisson; Number of chronic drugs at follow-up, adjusted for baseline value; Incidence Rate Ratio = 1.019, 95% CI 2-sided [0.833 to 1.246]

5. Secondary Outcome: Number of New Drugs Prescribed as a Result of the Intervention
Description: This outcome was not analysed
Time Frame: 4 months
Population: This outcome was not analyzed, as the drugs newly prescribed as a result of the intervention could not be distinguished from the other drugs newly prescribed.
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Health-related Quality of Life
Description: The EuroQol 5-Dimensions 5-Levels (EQ-5D-5L) tool was used to assess quality of life; this tool includes
  * a visual analog scale, ranging from 0 to 100, 100 indicating "the best health you can imagine" and 0 "the worst health you can imagine". Higher results indicate an higher quality of life.
  * 5 questions, each with 5 possible answers. Using a valuation set, the answers to individual questions were transformed in a numeric index value for each participants, with a maximum of 1 and an infinitely low minimum. Higher values indicates higher perceived health-related quality of life.
Time Frame: 4 months
Population: Data on this outcome were missing for some participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 26 | 25
units on a scale
  EQ-5D-5L scale | 63.5 (17.2) | 65.4 (22.4)
  EQ-5D-l index | 0.51 (0.31) | 0.61 (0.33)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Analysis for the scale component; Test type: Superiority; p = 0.769, Regression, Linear; Scale value at follow-up, adjusted for baseline value; Slope = -1.36, 95% CI 2-sided [-10.60 to 7.89]
Statistical Analysis 2: Comparison: Individual Deprescribing Intervention vs Control; Analysis for the index component; Test type: Superiority; p = 0.075, Regression, Linear; Scale value at follow-up, adjusted for baseline value; Slope = -0.096, 95% CI 2-sided [-0.202 to 0.01]

7. Secondary Outcome: Number of Common Drug-related Complaints at Follow-up
Description: Number of common drug-related complaints at follow-up
Time Frame: 4 months
Population: Data on this outcome at follow-up were missing for some participants, because of death or hospitalisation.
Measure: Mean (Standard Deviation); unit: Number of complaints
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 26 | 25
Number of complaints | 2.35 (2.60) | 1.44 (1.26)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.212, Mixed-effect regression, Poisson; Number at follow-up, adjusted for baseline value; Incidence Rate Ratio = 1.237, 95% CI 2-sided [0.886 to 1.727]

8. Other Pre Specified Outcome: Number of Deaths
Description: Number of deaths
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
Participants | 4 | 2
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.675, Fisher Exact; p-value = 0.675

9. Other Pre Specified Outcome: Number of Participants Hospitalized
Description: Number of participants hospitalized at any time during the study
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
Participants | 3 | 1
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.615, Fisher Exact; p-value = 0.615

10. Other Pre Specified Outcome: Days Spent in Hospital
Description: Average number of days spent in hospital during the study period
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
Number of days | 3.6 (15.8) | 0.6 (2.9)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.366, Wilcoxon (Mann-Whitney); p-value = 0.366

11. Other Pre Specified Outcome: Number of Falls Per Participant
Description: Average number of falls during the study period
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: falls
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
falls | 0.45 (0.89) | 0.48 (0.80)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.738, Wilcoxon (Mann-Whitney); p-value = 0.738

12. Other Pre Specified Outcome: Number of Participants Who Fell
Description: Number of participants who fell at least once during the study period
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
Participants | 9 | 9
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.781, Wilcoxon (Mann-Whitney); p-value = 0.781

13. Other Pre Specified Outcome: Number of Falls in Participants That Fell at Least Once
Time Frame: 4 months
Population: Only the participants who fell at least once were included in this analysis
Measure: Mean (Standard Deviation); unit: Number of falls
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 9 | 9
Number of falls | 1.6 (1.0) | 1.4 (0.7)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.958, Fisher Exact; p-value = 0.958

14. Other Pre Specified Outcome: Number of Days Spent With Physical Restraints
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Individual Deprescribing Intervention | Control
Number analyzed (Participants) | 31 | 27
days | 15.6 (39.1) | 15.1 (39.1)
Statistical Analysis 1: Comparison: Individual Deprescribing Intervention vs Control; Test type: Superiority; p = 0.911, Wilcoxon (Mann-Whitney); p-value = 0.911

ADVERSE EVENTS:
Time Frame: 4 months
Description: Adverse events were collected for the intervention group only.
Groups:
- 0.911 0.911 Individual Deprescribing Intervention: Participants allocated to the intervention arm will receive the Individual Deprescribing Intervention (pharmacist-led medication review, followed by the creation of a deprescribing plan by the pharmacist, physician and responsible nurse).
  Individual Deprescribing Intervention: The pharmacist responsible for the nursing home will perform a medication review (type 3). The results of this review will be discussed with the physician and nurse responsible for this participant, with the goal of creating a personalised deprescribing plan. Once validated by the physician, this plan will be submitted to the participant for approval.
Arm/Group | 0.911 0.911 Individual Deprescribing Intervention | Control
All-Cause Mortality (participants affected / at risk) | 5/32 | 4/30
Serious Adverse Events (participants affected / at risk) | 4/31 | 0/0
Other Adverse Events (participants affected / at risk) | 0/31 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.911 0.911 Individual Deprescribing Intervention (N=31) | Control (N=0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gout crisis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oedema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03655405/Prot_SAP_000.pdf